CLINICAL TRIAL: NCT02703961
Title: Multicenter Study on Efficacy and Safety of Concurrent and Adjuvant Chemotherapy With Cisplatin and Docetaxel Combined With Radiotherapy for Local Advanced Cervical Cancer
Brief Title: Randomized Control Trial on Efficacy and Safety of Concurrent and Adjuvant Chemotherapy for the Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Mei Shi, chair of department, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJFL-2016-02-LACC-TP triweekly
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Cervical Cancer
Keywords: CCRT; adjuvant chemotherapy; cisplatin and docetaxel
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Docetaxel; Brachytherapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental (Experimental): concurrent and adjuvant chemotherapy with cisplatin and docetaxel combined radical radiotherapy.
  During external beam radiotherapy: cisplatin 60mg/m2, d1,d22; docetaxel 60mg/m2, d1,d22.
  After external beam radiotherapy: cisplatin 75mg/m2, d43,d64;
  The patients also undergo external-beam radiation therapy once daily, 5 days a week, for approximately 5 weeks. Patients then undergo high-dose rate intracavitary brachytherapy.
  docetaxel 75mg/m2, d43,d64.
  Interventions: Drug: concurrent chemotherapy with cisplatin; Drug: concurrent chemotherapy with docetaxel; Radiation: pelvic radiotherapy; Radiation: brachytherapy; Drug: adjuvant chemotherapy with cisplatin and docetaxel
- control (Other): standard chemoradiotherapy with weekly cisplatin.
  Patients receive cisplatin IV over 60-90 minutes on days 1, 8, 15, 22, and 29.
  Patients also undergo external-beam radiation therapy once daily, 5 days a week, for approximately 5 weeks. Patients then undergo high-dose rate intracavitary brachytherapy.
  Interventions: Drug: concurrent chemotherapy with cisplatin; Radiation: pelvic radiotherapy; Radiation: brachytherapy

INTERVENTIONS:
Drug: concurrent chemotherapy with cisplatin — in experimental group: cisplatin 60mg/m2, d1,d22;
  Other Names: cisplatin
Drug: concurrent chemotherapy with docetaxel — in experimental group: docetaxel 60mg/m2, d1,d22;
  Other Names: docetaxel
  Arms: experimental
Radiation: pelvic radiotherapy — external beam radiotherapy for whole pelvix with 50Gy/25f boost radiotherapy for pelvic lymph node metastasis with 12-14Gy/4-7f.
  Other Names: external beam radiotherapy
Radiation: brachytherapy — CT/MRI guided brachytherapy or x-ray guided brachytherapy
Drug: adjuvant chemotherapy with cisplatin and docetaxel — cisplatin 75mg/m2, d43,d64; docetaxel 75mg/m2, d43,d64
  Arms: experimental

SUMMARY:
The standard treatment of local advanced cervical cancer is concurrent chemoradiotherapy. The 3 year disease free survival was about 50-70%. The distant metastasis is the main cause of failure in local advanced cervical cancer treated with 3-dimensional conformal radiotherapy (3D-CRT) or intensity modulated radiotherapy (IMRT). The purpose of this study is to investigate the efficacy and tolerance of concurrent and adjuvant chemotherapy with cisplatin and docetaxel for local advanced cervical cancer. It was expected that the 3 year disease free survival would be increased by 10% with this new treatment schedule.

DETAILED DESCRIPTION:
The cervical cancer is the most common malignant gynecological tumor in the developing area. From 1999, the concurrent chemoradiotherapy has been established as the standard treatment for local advanced cervical cancer. The modern radiotherapy techniques, such as 3 dimensional conformal radiotherapy(3D-CRT), intensity modulated radiotherapy(IMRT), image guided 3-dimensional brachytherapy(3D-BT), was widely used for the treatment of cervical cancer. The recently clinical outcome showed that the 3 year local and regional control was more than 90%［1-3］. The distant metastasis has proved to be the main cause of failure and death, especially for the patient with pelvic lymph node metastasis, large volume of tumor and advanced FIGO stage. the data showed that the 3 year distant metastasis free survival and overall survival were 64.7% and 64.6% respectively for the patient with huge pelvic lymph node metastasis and FIGO stage III- IVA. The system treatment pointing at the distant metastasis has become to be the topic of clinical investigation.

Dueñas-González A'［4］ study demonstrated that the 3 year progress free survival and distant metastasis free survival has increased by 8.9% and 8.3% by the radial radiotherapy combined with concurrent chemotherapy with weekly gemcitabine and cisplatin and adjuvant chemotherapy with triweekly gemcitabine and cisplatin. Ryu SY［5］ also reported the triweekly concurrent cisplatin with 3 cycles improved survival outcomes compared with weekly concurrent cisplatin. Retrospective studies by Tang and Jelavić-TB［6-7］ suggested that the adjubant chemotherapy after CCRT has better DMFS and OS.

The aim of present study is to prospectively investigate the efficacy and safety of concurrent and adjuvant chemotherapy with cisplatin and docetaxel for patients with local advanced cervical cancer, especially for those with FIGO III-IVA with or without pelvic lymph node metastasis and the FIGO IB2-IIB with pelvic lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven, invasive squamous cell carcinoma, adenocarcinoma, or adenosquamouscarcinoma of the cervix
2. FIGO clinical stage IB2-IIB with pelvic lymph node metastasis or FIGO clinical stage III-IVA with or without pelvic lymph node metastasis
3. ECOG performance score 0-1
4. The bone marrow, hepatic and renal function was normal at registration
5. The patients signed informed consent

Exclusion Criteria:

1. clear cell and small cell neuroendocrine, sarcoma
2. FIGO stage IVB
3. Prior invasive malignancy
4. Prior systemic chemotherapy
5. Prior radiotherapy to the pelvis or abdomen
6. Severe, active co-morbidity
7. Women who are pregnant
8. immunocompromised status

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 598 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 year

SECONDARY OUTCOMES:
overall survival | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: mei shi, professor, Principal Investigator — Xijing Hospital, the Fourth Military Medical University
Locations (3):
- China (3):
  - Xijing hospital, the Fourth Military Medical University, Xi'an, Shaanxi
  - Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University, Xi’an, Shanxi
  - Department of Radiation Oncology, Xijing Hospital, Fourth Military, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Jelavic TB, Mise BP, Strikic A, Ban M, Vrdoljak E. Adjuvant Chemotherapy in Locally Advanced Cervical Cancer After Treatment with Concomitant Chemoradiotherapy--Room for Improvement? Anticancer Res. 2015 Jul;35(7):4161-5. PMID 26124372
- [Result] Tharavichitkul E, Chakrabandhu S, Wanwilairat S, Tippanya D, Nobnop W, Pukanhaphan N, Galalae RM, Chitapanarux I. Intermediate-term results of image-guided brachytherapy and high-technology external beam radiotherapy in cervical cancer: Chiang Mai University experience. Gynecol Oncol. 2013 Jul;130(1):81-5. doi: 10.1016/j.ygyno.2013.04.018. Epub 2013 Apr 17. PMID 23603369
- [Result] Gill BS, Kim H, Houser CJ, Kelley JL, Sukumvanich P, Edwards RP, Comerci JT, Olawaiye AB, Huang M, Courtney-Brooks M, Beriwal S. MRI-guided high-dose-rate intracavitary brachytherapy for treatment of cervical cancer: the University of Pittsburgh experience. Int J Radiat Oncol Biol Phys. 2015 Mar 1;91(3):540-7. doi: 10.1016/j.ijrobp.2014.10.053. Epub 2015 Jan 30. PMID 25680598
- [Result] Tinkle CL, Weinberg V, Chen LM, Littell R, Cunha JAM, Sethi RA, Chan JK, Hsu IC. Inverse Planned High-Dose-Rate Brachytherapy for Locoregionally Advanced Cervical Cancer: 4-Year Outcomes. Int J Radiat Oncol Biol Phys. 2015 Aug 1;92(5):1093-1100. doi: 10.1016/j.ijrobp.2015.04.018. Epub 2015 Jul 14. PMID 26194683
- [Result] Duenas-Gonzalez A, Zarba JJ, Patel F, Alcedo JC, Beslija S, Casanova L, Pattaranutaporn P, Hameed S, Blair JM, Barraclough H, Orlando M. Phase III, open-label, randomized study comparing concurrent gemcitabine plus cisplatin and radiation followed by adjuvant gemcitabine and cisplatin versus concurrent cisplatin and radiation in patients with stage IIB to IVA carcinoma of the cervix. J Clin Oncol. 2011 May 1;29(13):1678-85. doi: 10.1200/JCO.2009.25.9663. Epub 2011 Mar 28. PMID 21444871
- [Result] Ryu SY, Lee WM, Kim K, Park SI, Kim BJ, Kim MH, Choi SC, Cho CK, Nam BH, Lee ED. Randomized clinical trial of weekly vs. triweekly cisplatin-based chemotherapy concurrent with radiotherapy in the treatment of locally advanced cervical cancer. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e577-81. doi: 10.1016/j.ijrobp.2011.05.002. Epub 2011 Aug 11. PMID 21840137
- [Result] Tang J, Tang Y, Yang J, Huang S. Chemoradiation and adjuvant chemotherapy in advanced cervical adenocarcinoma. Gynecol Oncol. 2012 May;125(2):297-302. doi: 10.1016/j.ygyno.2012.01.033. Epub 2012 Jan 31. PMID 22307061